CLINICAL TRIAL: NCT06637904
Title: TriVerity™ for Improved Management of Emergency Department (ED) Patients With Suspected Infections
Acronym: TIMED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inflammatix (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: INF-29
Record Dates: First submitted 2024-09-05; First posted 2024-10-15 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Sepsis; Infections; Tachycardia; Fever
MeSH Terms: conditions — Sepsis; Infections; Tachycardia; Fever

STUDY DESIGN:
Intervention Model Description: Pre-phase is the control arm and Post-phase is the interventional arm (uses TriVerity Test intervention)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Pre-phase standard of care (No Intervention): Participants in the pre-phase, treated with standard of care, will be gathered from a retrospective database using propensity matching.
- Post-phase TriVerity Test (Experimental): Participants in the post-phase will be managed incorporating the TriVerity Test results with standardized guidance for interpretation and resulting management actions.
  Interventions: Diagnostic Test: TriVerity Test

INTERVENTIONS:
Diagnostic Test: TriVerity Test — Participants in the post-phase of the study will have a 2.5 ml whole blood draw obtained via venipuncture into a PAXgene® Blood RNA tube. Blood samples will be processed using the TriVerity Cartridge on the Myrna Instrument located in the ED.
  Arms: Post-phase TriVerity Test

SUMMARY:
A pre/post interventional use trial, with ED patients who are initially triaged to locations other than a dedicated patient room in the main ED (e.g., waiting room, hallway bed, and/or the staging area/fast track area) with suspected infection and tachycardia or fever will be enrolled. Study conduct will be performed under an Investigational Device Exemption (IDE) from the Food and Drug Administration (FDA). Participants in the pre-phase, treated with standard of care, will be gathered from a retrospective database using propensity matching, whereas participants in the post-phase will be managed incorporating the TriVerity™ Acute Infection and Sepsis Test results with standardized guidance for interpretation and resulting management actions. Many outcomes will be captured and compared between the pre- and post-phase phases including sepsis bundle compliance, patient disposition, appropriate use of antimicrobials (antibiotics and antivirals) and health economic findings. Safety measures for participants in the post-phase will include patient follow-up at predefined time points. The objective is to demonstrate improvement of patient management when incorporating the TriVerity Test result compared to standard of care. Improvements based on diagnostic (bacterial vs viral vs non-infectious inflammation) and prognostic (need for 7-day ICU level care) readouts of the TriVerity Test result will be tracked.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Participant presents to ED with ALL of the below:

   2.1. Suspected acute infection (e.g., respiratory, urinary, abdominal, skin & soft-tissue infection, meningitis/encephalitis, or any other infection), and 2.2. Either heart rate >100 beats per minute or/and temperature >38C. 2.3. NOT immediately roomed in a primary designated treatment location,( i.e., they can be in the waiting room, ED triage hallways, and/or ED staging area/fast track area).
3. Able to provide informed consent, or consent by legally authorized representative.
4. Reachable via confirmed working cell phone (with backup contact number) and willing to respond to follow-up safety checks (see below for details).

Exclusion Criteria:

1. Patient-reported treatment with systemic antibiotics, systemic antiviral agents or systemic antifungal agents within the past 7 days prior to presentation in the waiting room of the ED. Participants will not be excluded for use of:

   1. Antiviral treatment for chronic viral infections, i.e., HIV, hepatitis B and hepatitis C
   2. Topical antibiotics, topical antivirals or topical antifungal agents
   3. Anti-herpes prophylaxis aiding suppression of a recuring herpes infection
   4. Single dose of one or combination of peri-operative (prophylactic) antibiotics
2. Patients receiving palliative or hospice care, or those receiving limited interventional care (see Appendix B).
3. Prisoners, mentally disabled, or unable to give consent. Should the patient not be able to provide informed consent the legally authorized representative can provide the consent on behalf of the patient.
4. Participants receiving experimental therapy or already enrolled in an interventional clinical trial in which a subject receives some type of intervention, which can include but is not limited to investigational drugs, medical devices, or vaccines. Participants that are enrolled in non-interventional or observational clinical trials will be allowed to participate in this clinical trial.
5. Participants previously enrolled in the present clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
SEP-1 bundle compliance | Within 72 hours of ED admission
  Mandatory hospital procedures for patients admitted with suspected sepsis
Time to final ED disposition order | Date of enrollment (Day 0) to final Follow Up call (up to 35 days)
  Time from Triage (on Day 0) to the Time the ED physician orders the subject disposition (i.e., where the subject will go next: admittance or discharge).

SECONDARY OUTCOMES:
Percent of patients with antibiotics given in the ED combined with noninferior safety outcomes | Date of enrollment (Day 0) to final Follow Up call (up to 35 days)
  Calculated based on number of patients given antibiotics in ED
Emergency Department LOS | Date of enrollment (Day 0) to final Follow Up call (up to 35 days)
  Length of Stay
Diagnostic ordering practices | Date of enrollment (Day 0) to 72 hours
  Capturing the diagnostic ordering practices of attending physician (comparing physician choices and decisions before and after the TriVerity Test)
Hospital admission rates | Date of enrollment (Day 0) to 72 hours
  Overall admission rates for patients that meet study criteria from emergency department to other location (e.g., ICU)
Total hospital costs | Date of enrollment (Day 0) to 28 days
  Overall hospital costs for patients that meet study criteria

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - OSF HealthCare Saint Francis Medical Center, Peoria, Illinois
  - Johns Hopkins Department of Emergency Medicine, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No